CLINICAL TRIAL: NCT06664957
Title: The Role of the Antioxidant Effects of Vitamin C in Improving the Prognosis of Patients With Chronic Obstructive Pulmonary Disease: A Multicenter, Randomized, Double-Blind, Parallel-Group, Placebo-Controlled Study.
Brief Title: Vitamin C's Antioxidant Effects and COPD Prognosis
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-R064-02
Record Dates: First submitted 2024-10-27; First posted 2024-10-30 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: COPD (Chronic Obstructive Pulmonary Disease)
Keywords: Vitamin C; Antioxidant Effects; Prognosis
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin C group (Experimental): Participants in this group will receive 400 mg of a nutrient supplement (Vitamin C) daily, administered as two 100 mg tablets in the morning and two 100 mg tablets in the evening for 12 months. Vitamin C is provided as a dietary supplement with the goal of supporting antioxidant defense, potentially reducing oxidative stress and improving clinical outcomes in COPD patients. Regular follow-ups will occur every 3 months to monitor exacerbations, quality of life, and safety.
  Interventions: Dietary Supplement: Vitamin C (Ascorbic Acid)
- Placebo group (Placebo Comparator): Participants in this group will receive a matching placebo, administered as two tablets in the morning and two tablets in the evening for 12 months. The placebo is identical in appearance to the Vitamin C supplement but contains no active ingredients. Follow-up visits will occur every 3 months, identical to the Vitamin C group, to monitor clinical outcomes, quality of life, and safety.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin C (Ascorbic Acid) — Participants in this arm will receive 400 mg of Vitamin C, administered as two 100 mg tablets in the morning and two 100 mg tablets in the evening, for a total of 12 months. The intervention aims to support antioxidant defense and improve clinical outcomes in COPD patients.
  Arms: Vitamin C group
Other: Placebo — Participants in this group will receive a placebo, identical in appearance to the active nutrient supplement (Vitamin C) tablets, with no active ingredients. The placebo will be administered as two tablets in the morning and two tablets in the evening (four tablets per day) for a duration of 12 months, serving as a control to compare the effects of the active intervention.
  Arms: Placebo group

SUMMARY:
This multicenter, randomized, double-blind, placebo-controlled clinical trial aims to evaluate the efficacy of Vitamin C supplementation in improving the prognosis of patients with Chronic Obstructive Pulmonary Disease (COPD) through its antioxidant effects.

The primary objectives of the study are to determine:

1. Whether Vitamin C reduces the frequency of acute COPD exacerbations.
2. Whether Vitamin C improves pulmonary function and health-related quality of life in patients with COPD.

The study will compare Vitamin C to a placebo to assess its impact on oxidative stress and its potential to enhance clinical outcomes in COPD management.

Participants will:

1. Receive either daily oral Vitamin C supplementation or a placebo for a period of 6 months. Undergo monthly clinical evaluations, including spirometry and symptom assessments.
2. Report any adverse events or health changes during the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Age 40-80 years (including 40 and 80).
2. Patients with COPD classified as GOLD stages 2-4:

   Post-bronchodilator FEV1/FVC < 70% and FEV1 < 80% of predicted value.
3. No respiratory infection or acute exacerbation of COPD within 4 weeks prior to enrollment. Acute exacerbation is defined as an acute worsening of respiratory symptoms requiring additional treatment.
4. The patient voluntarily consents to participate in the study, is capable of verbal or written communication, and can understand and sign the informed consent form. The patient must also be able to complete the necessary assessments required for the study.

Exclusion Criteria:

1. Presence of other respiratory diseases such as alpha-1 antitrypsin deficiency, primary ciliary dyskinesia, active pulmonary infection (e.g., tuberculosis), lung cancer, pulmonary fibrosis, cystic fibrosis, obesity hypoventilation syndrome, sarcoidosis, pulmonary hypertension, or clinically significant interstitial lung disease (patients with COPD as the primary disease and comorbid bronchiectasis may be included).
2. History of asthma or asthma-COPD overlap syndrome: Patients currently diagnosed with asthma, according to GINA or other recognized guidelines, will be excluded. Patients with a childhood history of asthma (defined as diagnosis before age 18 and fully resolved) may be included.
3. History of lung resection or expected need for lung volume reduction surgery during the study.
4. Clinically significant abnormalities on chest CT that are not attributable to COPD.
5. Presence of clinically significant cardiovascular, neurological, psychiatric, renal, hepatic, immunological, gastrointestinal, genitourinary, musculoskeletal, dermatological, sensory, endocrine diseases, or hematological abnormalities, as judged by the investigator, that may affect patient safety or confound the effectiveness or safety analysis during the study.
6. Unstable cardiac disease: Patients will be excluded if they have any of the following conditions: a. Myocardial infarction, unstable angina/acute coronary syndrome, coronary artery bypass graft (CABG) surgery, or percutaneous coronary intervention (PCI) within the past 6 months. b. Structural heart disease such as hypertrophic cardiomyopathy or significant valvular disease. c. Unstable or life-threatening arrhythmias requiring intervention within the past 3 months. d. NYHA class II-IV heart failure.
7. Active malignancy: Patients with active cancer will be excluded.
8. Recent Vitamin C use: Patients who have used Vitamin C supplements within the last 4 weeks will be excluded.
9. Diabetes: Patients with poorly controlled diabetes or fasting blood glucose > 10 mmol/L will be excluded.
10. History of kidney stones or diagnosis of kidney stones within the past year, as high doses of Vitamin C may increase the risk of stone formation.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 650 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Annual Exacerbation Rate | 12 months
  Annual exacerbation rate will be measured as the total number of acute exacerbations of COPD experienced by each patient during the 12-month follow-up period. An exacerbation is defined as a worsening of COPD symptoms requiring additional treatment or hospitalization.

SECONDARY OUTCOMES:
Time to First Exacerbation | 3 months, 6 months, 9 months, 12 months
  Time from randomization to the first acute exacerbation of COPD requiring additional treatment or hospitalization.
Frequent Exacerbations (≥2 Events/Year) | 12 months
  The number of patients experiencing two or more acute exacerbations of COPD during the 12-month follow-up period.
Moderate to Severe COPD Exacerbations | 12 months
  The total number of moderate to severe COPD exacerbations, defined by the need for systemic corticosteroids, antibiotics, or hospitalization.
Change in the Average Daily Puffs of Rescue Medication | Baseline, 3 months, 6 months, 9 months, 12 months
  This outcome measure assesses the change from baseline in the average number of daily puffs of rescue medication (e.g., short-acting bronchodilators) used by participants. It serves as an indicator of changes in symptom control and the need for immediate symptom relief throughout the study duration.
Change in COPD Assessment Test (CAT) Score | Baseline, 3 months, 6 months, 9 months, 12 months
  Assesses the longitudinal change in COPD Assessment Test (CAT) score from baseline, an 8-item patient-reported outcome measure evaluating the impact of COPD on health status. The CAT score ranges from 0 to 40, with higher scores reflecting a more significant health impact and symptom burden due to COPD.
Change in St. George's Respiratory Questionnaire (SGRQ) Score | Baseline, 3 months, 6 months, 9 months, 12 months
  Measures the change in total score from baseline on the St. George's Respiratory Questionnaire (SGRQ), a validated health-related quality of life assessment specific to respiratory diseases. The SGRQ score ranges from 0 to 100, where higher scores denote poorer health-related quality of life and greater disease impact.
Change in Hospital Anxiety and Depression Scale (HADS) Score | Baseline, 3 months, 6 months, 9 months, 12 months
  Evaluates the change from baseline in Hospital Anxiety and Depression Scale (HADS) score. The HADS comprises two 7-item subscales that independently assess anxiety and depression, each subscale scored from 0 to 21. Higher scores on either subscale indicate more severe symptoms of anxiety or depression.
Mortality (All-Cause, Cardiovascular, Respiratory) | 3 months, 6 months, 9 months, 12 months
  All-cause mortality, cardiovascular mortality, and respiratory system mortality during the study period.
Adverse Events (AEs) and Serious Adverse Events (SAEs) | 3 months, 6 months, 9 months, 12 months
  The safety of Vitamin C supplementation will be evaluated by monitoring the incidence and severity of adverse events (AEs) and serious adverse events (SAEs), as well as any abnormal laboratory findings. This includes tracking any unexpected health outcomes or complications that may arise during the study.
Proportion of Days without Rescue Medication Use | Baseline, 3 months, 6 months, 9 months, 12 months
  This outcome measure calculates the proportion of days during the 12-month follow-up period on which participants did not require rescue medication. It reflects the frequency of stable symptom control, with fewer acute episodes necessitating immediate relief.
Number of Emergency Visits due to COPD Exacerbations | 3 months, 6 months, 9 months, and 12 months
  This outcome measure records the number of emergency visits required due to COPD exacerbations over the study period.
Number of Hospitalizations due to COPD Exacerbations | 3 months, 6 months, 9 months, and 12 months
  This outcome measure records the number of hospital admissions required due to COPD exacerbations.
Length of Hospital Stay | 3 months, 6 months, 9 months, and 12 months
  This outcome measure evaluates the duration of hospital stay (in days) following hospitalization for COPD exacerbations.

IPD SHARING:
Plan to Share IPD: No